CLINICAL TRIAL: NCT05420389
Title: Breast Massage and Hot Compress Application to Mothers With Premature Babies at Newborn Intensive Care University Effect on Milk Release and Anxiety: Randomized Controlled Study
Brief Title: Breast Massage and Hot Compress Application to Mothers With Premature Babies at Newborn Intensive Care University Effect on Milk Release and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seyma Ertugral (Other)
Responsible Party: Sponsor-Investigator, Seyma Ertugral, Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: gülhane sbu
Record Dates: First submitted 2022-04-23; First posted 2022-06-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Breast Milk Collection; Breast Pumping; Massage Therapy
Keywords: Breast Milk; Premature; Milking Pump; Hot Compress; Breast Massage; Anxiety; randomized controlled study
MeSH Terms: conditions — Breast Milk Expression; Premature Birth; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There will be 4 groups.three interventional and one control group.
Who Masked: Participant
Masking Description: The volunteer who is in the latent phase of labor will not know which group she will be in before joining the study. After accepting to participate in the study, the volunteer will be informed about which group she will be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- breast massage (Experimental): The mothers who were included in the breast massage group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the state anxiety scale were filled out on the first day. These mothers were shown breast massage during the use of milking pumps, they were provided with their own application and a brochure was given explaining the application.As long as the breast milk follow-up form to record the amounts of milk they milked was in the hospital, the researcher explained how to fill it out when discharged and was asked to fill out the last-day state anxiety scale (SATI-I). Milk amounts are measured in ml.
  Interventions: Other: breast massage
- hot compress (Experimental): Mothers who were included in the hot application group were informed about the use of milking pumps in the routine application of the hospital and the state anxiety scale (STAI-I) was filled out on the first day. These mothers were shown the hot application they would make during the use of milking pumps, they were provided with the application and a brochure was given explaining the application.The hot chest compress to be used in this group will be used in the Lansinoh brand Thera°Pearl® Hot Breast Therapy pad, which is sold in medical medicines in pharmacies approved by the Ministry of Health.The breast milk follow-up form, in which they will record the amounts of milk they milk, was explained by the researcher in the hospital and how to fill it out when they were discharged, and they were asked to fill out a last-day anxiety scale.
  Interventions: Other: hot compress
- breast massage-hot compress (Experimental): Mothers who were included in the breast massage and hot application group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the state anxiety scale were filled out on the first day. These mothers were shown breast massage and hot application during the use of milking pumps, they were provided with their own application and a brochure was given explaining the application.The breast milk follow-up form, in which they will record the amounts of milk they milk, was explained by the researcher in the hospital and how to fill it out when they were discharged, and they were asked to fill out a last-day anxiety scale.
  Interventions: Other: breast massage-hot compress
- control group (No Intervention): The mothers who were included in the control group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the state anxiety scale were filled out on the first day. These mothers were told by the researcher how to fill out the breast milk follow-up form for 4 days as long as they were in the hospital. Milk amounts are measured in ml. On the last day, the state anxiety scale has been filled.

INTERVENTIONS:
Other: breast massage — Mothers who were included in the breast massage group who met the research criteria were informed about the use of milking pumps in the routine application of the hospital and the condition anxiety scale was filled out on the first day. These mothers were shown breast massage during the use of milking pumps, they were provided with their own application and a brochure was given explaining the application.As long as the breast milk follow-up form to record the amounts of milk they milked was in the hospital, the researcher explained how to fill it out when discharged and was asked to fill out the last-day conditional anxiety scale (SATI-I). Milk amounts are measured in ml.
  Arms: breast massage
Other: hot compress — Mothers who were included in the hot application group were informed about the use of milking pumps in the routine application of the hospital and the condition anxiety scale (STAI-I) was filled out on the first day. These mothers were shown the hot application they would make during the use of milking pumps, they were provided with the application and a brochure was given explaining the application.The hot chest compress to be used in this group will be used in the Lansinoh brand Thera°Pearl® Hot Breast Therapy pad, which is sold in medical medicines in pharmacies approved by the Ministry of Health.The breast milk follow-up form, in which they will record the amounts of milk they milk, was explained by the researcher in the hospital and how to fill it out when they were discharged, and they were asked to fill out a last-day anxiety scale.
  Arms: hot compress
Other: breast massage-hot compress — Mothers who were included in the breast massage and hot application group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the condition anxiety scale were filled out on the first day. These mothers were shown breast massage and hot application during the use of milking pumps, they were provided with their own application and a brochure was given explaining the application.As long as the breast milk follow-up form to record the amounts of milk they milked was in the hospital, the researcher explained how to fill it out when discharged and was asked to fill out the last-day conditional anxiety scale (SATI-I). Milk amounts are measured in ml.
  Arms: breast massage-hot compress

SUMMARY:
This research was carried out in order to determine the effect of breast massage and hot compresses on milk release and anxiety to mothers with premature babies in YYBU (Neonatal Intensive Care Unit)

DETAILED DESCRIPTION:
Participants who met the criteria for inclusion of the study were informed about the purpose of the research, the scales used, the data to be collected and the purposes of use of this data. Participants who agreed to participate voluntarily in the study were given a questionnaire form in an environment where they could respond without distraction in their clinic and responded under the supervision of the researcher. The answer to the questionnaire was completed in approximately 10-15 minutes. Suitable for the research group in which participants are included; control group, breast massage application group, hot compress group to the breast, massage to the breast and data collection form suitable for hot compress group.Participants were followed by the post op 48 hour researcher. A mother with 120 premature babies who met the criteria for inclusion in the study was taken. The applications carried out in the study were shown to the mother by the researcher in a hands-on manner, explained and given a brochure explaining the application. The mothers who were included in the control group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the condition anxiety scale were filled out on the first day. These mothers were told by the researcher how to fill out the breast milk follow-up form for 4 days as long as they were in the hospital. Milk amounts are measured in ml. On the last day, the situation anxiety scale has been filled.

The mothers who were included in the breast massage group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the condition anxiety scale were filled out on the first day. These mothers were shown breast massage during the use of milking pumps, they were provided with a brochure explaining the application. As long as the breast milk follow-up form to record the amounts of milk they milked was in the hospital, the researcher explained how to fill it out when discharged and was asked to fill out the last-day conditional anxiety scale (SATI-I). Milk amounts are measured in ml.

Mothers who were included in the hot application group were informed about the use of milking pumps in the routine application of the hospital and the condition anxiety scale (STAI-I) was filled out on the first day. These mothers were shown the hot application they would make during the use of milking pumps, they were provided with the application and a brochure was given explaining the application.

The hot chest compress to be used in this group will be used in the Lansinoh brand Thera°Pearl® Hot Breast Therapy pad, which is sold in medical medicines in pharmacies approved by the Ministry of Health.

The breast milk follow-up form, in which they will record the amounts of milk they milk, was explained by the researcher in the hospital and how to fill it out when they were discharged, and they were asked to fill out a last-day anxiety scale. Mothers who were included in the breast massage and hot application group were informed about the use of milking pumps in the routine application of the hospital, the data collection form and the condition anxiety scale were filled out on the first day. These mothers were shown breast massage and hot application during the use of milking pumps, they were provided with their own application and a brochure was given explaining the application. The breast milk follow-up form, in which they will record the amounts of milk they milk, was explained by the researcher in the hospital and how to fill it out when they were discharged, and they were asked to fill out a last-day anxiety scale.

In the study, a MANDELA type milking pump was used, which belongs to the hospital where the work was carried out to milk the mothers. The milking pump setting of the mothers who participated in the study was also adjusted to moderate level.

Where the research was carried out : The research was carried out in the cesarean clinic of Ankara Etlik Zubeyde Women's Obstetrics and Gynecology Education and Research Hospital.

Universe and Sampling of The Research: The universe of this research is made up of patients who meet the criteria for inclusion in the cesarean clinic at Ankara Etlik Zubeyde Women's Obstetrics and Gynecology Education and Research Hospital and who agree to participate in the research. The sample size required for the research question created to examine the reduction of anxiety by increasing the amount of milk of the mother of breast massage, hot compress, breast massage-hot compress application to premature baby was examined in groups of thirtysomethings. Accordingly, the sample size of 120 people was grouped as Massage group [n=30], Hot group [n=30], Massage and Hot group [n=30] and Control group[n=30] as individuals. Randomization of groups was carried out through the computer randomization program Random Allocation Software program.

Data Evaluation: The analysis was conducted through the IBM SPSS Statistics 23 package program. When evaluating the study data, frequency (number, percentage) for categorical variables and descriptive statistics (mean, standard deviation, median, minimum, maximum) are given for numerical variables. The assumptions of normality of numerical variables by groups were examined by shapiro wilk normality test and it was observed that some variables were not distributed normally. Therefore, both parametric and non-parametric statistical methods were used in the study.The relationships between the two Independent categorical variables are interpreted by The Square analysis. Fisher Exact test results were used in cases where the expected value assumption was not provided in the Square analysis. The differences between more than two independent groups were looked at with the Kruskal Wallis test for variables that showed normal distribution, one-way variance analysis (ANOVA) for variables that did not have normal distribution. The differences between the Dependent Sample T Test and more than two dependent numeric variables for variables with normal distribution between two dependent numeric variables were examined with Friedman's Analysis.The power of the work is calculated by the GPower package program. In the study, the effect width was found to be 0.62 and the strength of the study, which was completed with a total of 120 people including 30 massages, 30 hot applications, 30 massages and hot treatments and 30 controls, was found to be 80.1% at the 0.05 significant level. Statistical signation was interpreted as 0.05 in the analysis.

Data Collection Tools:The research data were collected using the Data Collection Form, Spielberger's Situational Anxiety Inventory and Breast Milk Follow-up Form, which includes questions and sociodemographic data determined by the researchers in accordance with the subject of the research in line with the literature information.

ELIGIBILITY:
Inclusion Criteria:

* Who has agreed to participate in the research,
* Without communication barriers, She gave birth by C-section.

  * Preterm infant mothers who give birth before the 37th gestational week,
  * With a birth weight of less than 2000 grams,
  * Severely chronic disease, pregnancy complications or non-previous breast surgery,
  * Preterm infant mothers treated in YYBU will be included in the study.

Exclusion Criteria:

Failure to meet the inclusion criteria is the exclusion criteria.

Exclusion (Withdrawal) from the Study Criteria

* Failure to complete the data collection forms,
* the participant's desire to leave at any time of the study,
* the single-option information in the data collection forms,
* the failure to communicate with the mother after discharge in the collection of the work data.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 Years to 45 Years (Adult)
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Amount of Milk | Change from Amount of Milk 4 Days
  Milk quantities measured in ml.
Level of Anxiety | 1th day
  The state anxiety scale, the responses are classified as (1) Not at all, (2) A little, (3) A lot, and (4) Completely; Responses in the trait anxiety scale are classified as (1) almost never, (2) sometimes, (3) often, and (4) almost always. There are two kinds of statements (direct and reversed) in scales. While scoring these statements, those with a score of 1 turn into 4, and those with a score of 4 turn into 1. In direct statements, responses with a value of 4 indicate high anxiety. In reversed statements, responses with a value of 1 indicate high anxiety while those with a value of 4 indicate low anxiety. The scores obtained from both scales range from 20 to 80. The score obtained from the scales constitutes the individual's score to be interpreted at the level of anxiety. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Level of Anxiety | 4th day
  The state anxiety scale, the responses are classified as (1) Not at all, (2) A little, (3) A lot, and (4) Completely; Responses in the trait anxiety scale are classified as (1) almost never, (2) sometimes, (3) often, and (4) almost always. There are two kinds of statements (direct and reversed) in scales. While scoring these statements, those with a score of 1 turn into 4, and those with a score of 4 turn into 1. In direct statements, responses with a value of 4 indicate high anxiety. In reversed statements, responses with a value of 1 indicate high anxiety while those with a value of 4 indicate low anxiety. The scores obtained from both scales range from 20 to 80. The score obtained from the scales constitutes the individual's score to be interpreted at the level of anxiety. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Satisfaction Rating | 4th day
  Massage is a scale from 1 to 10 to determine the satisfaction of mothers from hot compresses, hot-massage compress applications. High score indicates satisfaction, low score indicates dissatisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik Zübeyde Hanım Kadın Hastalıkları Ve Doğum Hastanesi, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No